CLINICAL TRIAL: NCT02793661
Title: Study to Evaluate the Use of RenalGuard to Protect Patients at High Risk of AKI (STRENGTH)
Brief Title: Study to Evaluate the Use of RenalGuard to Protect Patients at High Risk of AKI
Acronym: STRENGTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Cardiovascular Research Center (Network)
Collaborators: RenalGuard Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REN-01
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Cardiovascular Disease; Acute Kidney Injury
MeSH Terms: conditions — Cardiovascular Diseases; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RenalGuard Arm (Experimental): In order to prevent patients from acute kidney injury, patients will receive the RenalGuard Therapy delivered by the RenalGuard system from one hour before the cardiovascular intervention to 4 hours after the intervention.
  Interventions: Device: RenalGuard
- Control Arm (Active Comparator): Patient will received standard treatment, as per ESC Guidelines 2014, to prevent from acute kidney injury.
  Interventions: Other: Control

INTERVENTIONS:
Device: RenalGuard — Replacement of urine output by infusion of a matched volume of sterile replacement solution to maintain a patient's intravascular fluid volume. Diuretic is administered to reach an optimum urine flow and protect efficiently the patients' kidneys.
  Arms: RenalGuard Arm
Other: Control — Hydration protocol following ESC Guidelines 2014
  Arms: Control Arm

SUMMARY:
The Strength study aim to evaluate the use of the RenalGuard device to protect the patients at high risk to develop acute kidney injury following a complex cardiovascular intervention requiring a high volume of contrast.

DETAILED DESCRIPTION:
The Strength Trial is a randomized, international (France and Germany) and multicentre (7) trial.

The patients population targeted is suffering from kidney insufficiency (estimated Glomerular Filtration Rate (eGFR) between 15 to 40 ml/min/m2) need to go through a complex cardiovascular intervention..

This is a population of patients at high risk to develop AKI following contrast media administration and complex cardiovascular interventions require a high amount of contrast.

Standard treatment is hydration but with risk of hyper and hypohydration for this population of patients. RenalGuard insure the replacement of the urine output by infusion of a matched volume of sterile replacement solution to maintain patients' intravascular fluid volume.

The patients are randomized to be protected from contrast-induced nephropathy with the use of RenalGuard or by standard hydration treatment and will be followed-up during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* 15 ml/min/m2 ≤ eGFR ≤ 40 ml/min/m2
* High volume contrast-requiring cardiovascular procedures (estimated contrast volume > 3 times eGFR value)
* Patient has agreed to all FU testing

Exclusion Criteria:

* Administration of iodine contrast media within 5 days before index procedure
* Emergency procedure or primary PCI
* Patients with pulmonary edema or cardiogenic shock (Killip 3 or 4)
* Hypoxemia defined as SaO2 ≤ 90% and/or PaO2 ≤ 80 mmHg on room air
* Acute Kidney Injury requiring dialysis before the procedure
* Multiple myeloma or cancer treated with chemotherapy
* Subjet is anuric
* Subject has been hospitalized for any change in renal function or has undergone renal replacement therapy (hemodialysis or hemofiltration) within the past month
* Known hypersensitivity to furosemide active ingredient or excipient
* Renal insufficiency with oligoanuria resistant to furosemide or caused by nephrotoxic or hepatotoxic substances
* Pre-coma or coma induced by an hepatic encephalopathy
* Severe hypokalemia, sever hyponatremia, hypovolemia with or without hypotension or dehydration
* Hypersensitivity to sulfamides
* Enrollment in another study unless the study is a registry or unless primary endpoint is reached
* Expected life expectancy < 1 year
* Pregnant or breastfeeding patient
* Patient under trusteeship or guardianship
* Patient is unable / unwilling to provide an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Occurence of contrast-induced nephropathy | Within 5 days
  The occurence of contrast-induced nephropathy will be determined:
  * by an elevation, within 3 days from requiring contrast-procedure, of the serum creatinine (rise of 0.3mg/dl or of 25% compared to basal value) and/or
  * by the need for dialysis within 5 fays from requiring contrast-procedure

SECONDARY OUTCOMES:
Change in serum creatinin value | at 12 +-1 months
Change in the estimated glomerular filtration rate | at 12 +-1 months
Percentage of patients on chronic dialysis | at 12 +-1 months
Percentage of patients on temporary dialysis | at 12 +-1 months
In hospital significant urinary bleeding, infection or any other major complication cause by the urinary catheter | within 5 days from procedure
Composite of major adverse cardiovascular and cerebrovascular events (death, myocardial infarction, stroke, revascularization) | at 12 +-1 months
Individual MACCEs components (death, myocardial infarction, stroke, revascularization) | at 12 +-1 months
Economic evaluation of RenalGuard compared to standard renal protection according to ESC guidelines | Index hospitalization (including staged procedures) and 12+- 1 months
  cost utility analysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Halpert, Study Director — RenalGuard Solutions, Inc.
Locations (7):
- France (4):
  - Hôpital Privé Jacques Cartier, Massy
  - Hôpital Privé Claude Galien, Quincy-sous-Sénart
  - CHU Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (3):
  - Universitätsklinikum Bonn, Bonn
  - Cardiovasculares Centrum Frankfurt, Frankfurt
  - St Josefs Hospital, Wiesbaden

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152